CLINICAL TRIAL: NCT04079322
Title: Fractional Iron Absorption in Response to an Acute Bout of Exercise
Brief Title: Iron Absorption and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Stephen R. Hennigar, Ph.D., Assistant Professor, Florida State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019.28633
Record Dates: First submitted 2019-08-12; First posted 2019-09-06 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): During the exercise arm, volunteers will complete a planned workout, as prescribed by the coach. The workout will be designed to be strenuous and induce an inflammatory response.
  Interventions: Other: Meal
- Rest (Experimental): The rest arm will be coordinated with a planned non-workout day, as prescribed by the coach, where volunteers are either scheduled to not run or go for an easy recovery run (<6 miles at a self-described "easy" pace) later in the afternoon.
  Interventions: Other: Meal

INTERVENTIONS:
Other: Meal — Participants will consume a meal containing a stable iron isotope following exercise or rest.

SUMMARY:
Iron is a nutritionally essential mineral required for optimal physical and cognitive performance. Endurance exercise often leads to declines in iron status; however, the reason for the decline is not known. The primary objective of the proposed study is to determine the effects of an acute bout of strenuous endurance exercise on iron absorption and status and markers of inflammation in human volunteers. The investigators hypothesize that an acute bout of strenuous endurance exercise, compared to rest, will reduce iron absorption, resulting in diminished iron status, and that reduced iron absorption will be negatively associated with markers of inflammation. A secondary objective is to monitor iron status throughout a season of competition.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Florida State University Cross Country team
* Refrain from using any pain-relievers (e.g., acetaminophen, nonsteroidal anti-inflammatory drugs such as aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product on the 2 study days
* Refrain from using vitamin or mineral supplements on the study days

Exclusion Criteria:

* Musculoskeletal injury that compromise the ability to exercise

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Change in fractional iron absorption | Red blood cells collected on day 0 and day 14
  Stable iron isotopes

SECONDARY OUTCOMES:
Change in concentration of ferritin in ng/mL | Day 0 and day 14
  Blood measure
Change in concentration of soluble transferrin receptor in nmol/L | Day 0 and day 14
  Blood measure
Change in concentration of hemoglobin in g/L | Day 0 and day 14
  Blood measure
Change in concentration of hematocrit as % | Day 0 and day 14
  Blood measure
Change in concentration of hepcidin in ng/mL | Day 0 and day 14
  Blood measure
Change in concentration of IL-6 in pg/mL | Day 0 and day 14
  Blood measure

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barney DE Jr, Cheung SN, Harris AR, Berryman CE, Hennigar SR. Dietary Intake and Diet Quality of Female and Male NCAA Division I Cross Country Runners from a Single University. Curr Dev Nutr. 2024 Oct 15;8(11):104475. doi: 10.1016/j.cdnut.2024.104475. eCollection 2024 Nov. PMID 39610765
- [Derived] Barney DE, Ippolito JR, Berryman CE, Hennigar SR. A Prolonged Bout of Running Increases Hepcidin and Decreases Dietary Iron Absorption in Trained Female and Male Runners. J Nutr. 2022 Sep 6;152(9):2039-2047. doi: 10.1093/jn/nxac129. PMID 35661896